CLINICAL TRIAL: NCT00467779
Title: A Phase 1 Dose-Escalation Study of the Safety and Pharmacokinetics of GDC-0973/XL518 Administered Orally Daily to Subjects With Solid Tumors
Brief Title: Study of Cobimetinib in Participants With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MEK4592g; GO01329 (Other: Hoffmann-La Roche); XL518-001 (Other: Exelixis)
Record Dates: First submitted 2007-04-18; First posted 2007-05-01 (Estimated); Results first posted 2016-07-22 (Estimated); Last update posted 2016-08-26 (Estimated); Status verified 2016-07

CONDITIONS: Solid Tumor
MeSH Terms: interventions — cobimetinib; Dextromethorphan; Midazolam

ARMS (5):
- Stage 1: Cobimetinib Dose Escalation (21/7 Schedule) (Experimental): Participants will receive cobimetinib (GDC-0973/XL518) at the starting dose of 0.05 mg/kg via solution or capsule, once daily for Days 1-21 of each 28-day cycle (21 days on drug followed by 7 days off treatment [21/7 schedule]). Treatment will continue until progressive disease (PD) or unacceptable toxicity for up to 1 year at the discretion of investigator and beyond 1 year with the agreement of the sponsor.
  Interventions: Drug: cobimetinib
- Stage 1A: Cobimetinib Dose Escalation (14/14 Schedule) (Experimental): Participants will receive cobimetinib at the starting dose of 60 mg via solution or capsule, once daily for Days 1-14 of each 28-day cycle (14 days on drug followed by 14 days off treatment [14/14 schedule]). Treatment will continue until progressive disease (PD) or unacceptable toxicity for up to 1 year at the discretion of investigator and beyond 1 year with the agreement of the sponsor.
  Interventions: Drug: cobimetinib
- Stage 2: Cobimetinib Expansion (21/7 Schedule) (Experimental): Participants will receive cobimetinib at the maximum tolerated dose (MTD) established in Stage 1, once daily for Days 1-21 of each 28-day cycle (21 days on drug followed by 7 days off treatment [21/7 schedule]). Treatment will continue until progressive disease (PD) or unacceptable toxicity for up to 1 year at the discretion of investigator and beyond 1 year with the agreement of the sponsor.
  Interventions: Drug: cobimetinib
- Stage 2 A: Cobimetinib Expansion (14/14 Schedule) (Experimental): Participants will receive cobimetinib at the MTD established in Stage 1A, once daily for Days 1-14 of each 28-day cycle (14 days on drug followed by 14 days off treatment [14/14 schedule]). Treatment will continue until progressive disease (PD) or unacceptable toxicity for up to 1 year at the discretion of investigator and beyond 1 year with the agreement of the sponsor.
  Interventions: Drug: cobimetinib
- Stage 3: Cobimetinib+Midazolam+Dextromethorphan (Experimental): Participants will receive a single dose of midazolam (2 mg of midazolam syrup) and dextromethorphan (30 mg tablet) on Cycle 1 Day 1, in the absence of cobimetinib. After a 2-day washout period, participants will receive 21 consecutive daily doses of cobimetinib (60-mg) followed by a 7-day washout period. Participants will receive another single dose of midazolam and dextromethorphan on Cycle 1 Day 15, in the presence of steady-state cobimetinib concentrations. In Cycle 2 and beyond participants will receive cobimetinib alone, administered as a 60-mg daily dose for 21 consecutive days in 28-day cycles (21/7 schedule).
  Interventions: Drug: cobimetinib; Drug: dextromethorphan; Drug: midazolam

INTERVENTIONS:
Drug: cobimetinib — Repeating oral dose
  Other Names: GDC-0973/XL518
Drug: dextromethorphan — In Stage III only: single dose of dextromethorphan
  Arms: Stage 3: Cobimetinib+Midazolam+Dextromethorphan
Drug: midazolam — In Stage III only: single dose of midazolam
  Arms: Stage 3: Cobimetinib+Midazolam+Dextromethorphan

SUMMARY:
This non-randomized, open-label, study will determine the highest safe dose of cobimetinib, how often it should be taken, how well participants with cancer tolerate cobimetinib and will assess the pharmacokinetic effect of midazolam and dextromethorphan on the study drug.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed solid tumor that is metastatic or unresectable, and for which standard curative or palliative measures do not exist or are no longer effective, and there are no known therapies to prolong survival
* Disease that is measurable according to Response Evaluation Criteria in Solid Tumors (RECIST)
* Adequate organ and marrow function
* Sexually active participants must use medically acceptable methods of contraception during the course of the study and at least 11 days after the last dose of study treatment
* Female participants of childbearing potential must have a negative serum pregnancy test at screening
* No other history of/or ongoing malignancy that would potentially interfere with the interpretation of the pharmacodynamic or efficacy assays

Exclusion Criteria:

* Anticancer treatment (e.g., chemotherapy, radiotherapy, cytokines, or hormones) within 28 days (6 weeks for nitrosoureas or mitomycin C, or 14 days for hormonal therapy or kinase inhibitors) before the first dose of study drug
* The participant has not recovered to Grade </=1 from adverse events (AEs) or to within 10% of baseline values due to investigational or other agents administered more than 28 days prior to study enrollment
* The participant has received another investigational agent within 28 days of the first dose of study drug
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, diabetes, symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia
* The participant is pregnant or breastfeeding
* The participant is known to be positive for the human immunodeficiency virus (HIV)
* Allergy or hypersensitivity to components of the cobimetinib formulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2007-05; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (4):
- United States (4):
  - Los Angeles, California
  - Stanford, California
  - Detroit, Michigan
  - Buffalo, New York

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study included following stages: Stage 1, Stage 1A, Stage 2, Stage 2A, and Stage 3. Different participants were recruited in each stage.
Groups:
- Stage 1 Cohort 01 - Cobimetinib 0.05 mg/kg (21/7): Participants received cobimetinib (GDC-0973/XL518) 0.05 milligrams per kilograms (mg/kg) via solution or capsule, once daily for Days 1-21 of each 28-day cycle (21 days on drug followed by 7 days off treatment [21/7 schedule]). Treatment was continued until progressive disease (PD) or unacceptable toxicity for up to 1 year at the discretion of investigator and beyond 1 year with the agreement of the sponsor.
- Stage 1 Cohort 02 - Cobimetinib 0.10 mg/kg (21/7): Participants received cobimetinib 0.10 mg/kg via solution or capsule, once daily for Days 1-21 of each 28-day cycle. Treatment was continued until PD or unacceptable toxicity for up to 1 year at the discretion of investigator and beyond 1 year with the agreement of the sponsor.
- Stage 1 Cohort 03 - Cobimetinib 0.20 mg/kg (21/7): Participants received cobimetinib 0.20 mg/kg via solution or capsule, once daily for Days 1-21 of each 28-day cycle. Treatment was continued until PD or unacceptable toxicity for up to 1 year at the discretion of investigator and beyond 1 year with the agreement of the sponsor.
- Stage 1 Cohort 04 - Cobimetinib 10 mg (21/7): Participants received cobimetinib 10 mg via solution or capsule, once daily for Days 1-21 of each 28-day cycle. Treatment was continued until PD or unacceptable toxicity for up to 1 year at the discretion of investigator and beyond 1 year with the agreement of the sponsor.
- Stage 1 Cohort 05 - Cobimetinib 20 mg (21/7): Participants received cobimetinib 20 mg via solution or capsule, once daily for Days 1-21 of each 28-day cycle. Treatment was continued until PD or unacceptable toxicity for up to 1 year at the discretion of investigator and beyond 1 year with the agreement of the sponsor.
- Stage 1 Cohort 06 - Cobimetinib 40 mg (21/7): Participants received cobimetinib 40 mg via solution or capsule, once daily for Days 1-21 of each 28-day cycle. Treatment was continued until PD or unacceptable toxicity for up to 1 year at the discretion of investigator and beyond 1 year with the agreement of the sponsor.
- Stage 1 Cohort 07 - Cobimetinib 60 mg (21/7); Stage 2 Cohort 20 - Cobimetinib 60 mg (Expansion) (21/7): Participants received cobimetinib 60 mg via solution or capsule, once daily for Days 1-21 of each 28-day cycle. Treatment was continued until PD or unacceptable toxicity for up to 1 year at the discretion of investigator and beyond 1 year with the agreement of the sponsor.
- Stage 1 Cohort 08 - Cobimetinib 80 mg (21/7): Participants received cobimetinib 80 mg via solution or capsule, once daily for Days 1-21 of each 28-day cycle. Treatment was continued until PD or unacceptable toxicity for up to 1 year at the discretion of investigator and beyond 1 year with the agreement of the sponsor.
- Stage 1A Cohort 01A - Cobimetinib 60 mg (14/14): Participants received cobimetinib 60 mg via solution or capsule, once daily for Days 1-14 of each 28-day cycle (14 days on drug followed by 14 days off treatment [14/14 schedule]). Treatment was continued until PD or unacceptable toxicity for up to 1 year at the discretion of investigator and beyond 1 year with the agreement of the sponsor.
- Stage 1A Cohort 02A - Cobimetinib 80 mg (14/14): Participants received cobimetinib 80 mg via solution or capsule, once daily for Days 1-14 of each 28-day cycle. Treatment was continued until PD or unacceptable toxicity for up to 1 year at the discretion of investigator and beyond 1 year with the agreement of the sponsor.
- Stage 1A Cohort 03A - Cobimetinib 100 mg (14/14); Stage 2A Cohort 30 - Cobimetinib 100 mg (Expansion) (14/14): Participants received cobimetinib 100 mg via solution or capsule, once daily for Days 1-14 of each 28-day cycle. Treatment was continued until PD or unacceptable toxicity for up to 1 year at the discretion of investigator and beyond 1 year with the agreement of the sponsor.
- Stage 1A Cohort 04A - Cobimetinib 125 mg (14/14): Participants received cobimetinib 125 mg via solution or capsule, once daily for Days 1-14 of each 28-day cycle. Treatment was continued until PD or unacceptable toxicity for up to 1 year at the discretion of investigator and beyond 1 year with the agreement of the sponsor.
- Stage 3 Cohort 40 - Cobimetinib+Midazolam+Dextromethorphan: Participants received a single dose of midazolam (2 mg of midazolam syrup) and dextromethorphan (30 mg tablet) on Cycle 1 Day 1, in the absence of cobimetinib. After a 2-day washout period, participants received 21 consecutive daily doses of cobimetinib (60-mg) followed by a 7-day washout period.Participants received another single dose of midazolam and dextromethorphan on Cycle 1 Day 15, in the presence of steady-state cobimetinib concentrations. In Cycle 2 and beyond received cobimetinib alone, administered as a 60-mg daily dose for 21 consecutive days in 28-day cycles.
Period: Stage 1
Arm/Group | Stage 1 Cohort 01 - Cobimetinib 0.05 mg/kg (21/7) | Stage 1 Cohort 02 - Cobimetinib 0.10 mg/kg (21/7) | Stage 1 Cohort 03 - Cobimetinib 0.20 mg/kg (21/7) | Stage 1 Cohort 04 - Cobimetinib 10 mg (21/7) | Stage 1 Cohort 05 - Cobimetinib 20 mg (21/7) | Stage 1 Cohort 06 - Cobimetinib 40 mg (21/7) | Stage 1 Cohort 07 - Cobimetinib 60 mg (21/7) | Stage 1 Cohort 08 - Cobimetinib 80 mg (21/7) | Stage 2 Cohort 20 - Cobimetinib 60 mg (Expansion) (21/7) | Stage 1A Cohort 01A - Cobimetinib 60 mg (14/14) | Stage 1A Cohort 02A - Cobimetinib 80 mg (14/14) | Stage 1A Cohort 03A - Cobimetinib 100 mg (14/14) | Stage 1A Cohort 04A - Cobimetinib 125 mg (14/14) | Stage 2A Cohort 30 - Cobimetinib 100 mg (Expansion) (14/14) | Stage 3 Cohort 40 - Cobimetinib+Midazolam+Dextromethorphan
Started | 4 | 3 | 3 | 3 | 3 | 6 | 7 | 7 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 4 | 3 | 3 | 3 | 3 | 5 | 7 | 7 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Disease Progression | 2 | 2 | 2 | 3 | 2 | 2 | 4 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Unspecified Reason | 1 | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Stage 1A
Arm/Group | Stage 1 Cohort 01 - Cobimetinib 0.05 mg/kg (21/7) | Stage 1 Cohort 02 - Cobimetinib 0.10 mg/kg (21/7) | Stage 1 Cohort 03 - Cobimetinib 0.20 mg/kg (21/7) | Stage 1 Cohort 04 - Cobimetinib 10 mg (21/7) | Stage 1 Cohort 05 - Cobimetinib 20 mg (21/7) | Stage 1 Cohort 06 - Cobimetinib 40 mg (21/7) | Stage 1 Cohort 07 - Cobimetinib 60 mg (21/7) | Stage 1 Cohort 08 - Cobimetinib 80 mg (21/7) | Stage 2 Cohort 20 - Cobimetinib 60 mg (Expansion) (21/7) | Stage 1A Cohort 01A - Cobimetinib 60 mg (14/14) | Stage 1A Cohort 02A - Cobimetinib 80 mg (14/14) | Stage 1A Cohort 03A - Cobimetinib 100 mg (14/14) | Stage 1A Cohort 04A - Cobimetinib 125 mg (14/14) | Stage 2A Cohort 30 - Cobimetinib 100 mg (Expansion) (14/14) | Stage 3 Cohort 40 - Cobimetinib+Midazolam+Dextromethorphan
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 8 | 6 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 8 | 6 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Not completed — Disease Progression | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 5 | 2 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0
Not completed — Unspecified Reason | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Period: Stage 2
Arm/Group | Stage 1 Cohort 01 - Cobimetinib 0.05 mg/kg (21/7) | Stage 1 Cohort 02 - Cobimetinib 0.10 mg/kg (21/7) | Stage 1 Cohort 03 - Cobimetinib 0.20 mg/kg (21/7) | Stage 1 Cohort 04 - Cobimetinib 10 mg (21/7) | Stage 1 Cohort 05 - Cobimetinib 20 mg (21/7) | Stage 1 Cohort 06 - Cobimetinib 40 mg (21/7) | Stage 1 Cohort 07 - Cobimetinib 60 mg (21/7) | Stage 1 Cohort 08 - Cobimetinib 80 mg (21/7) | Stage 2 Cohort 20 - Cobimetinib 60 mg (Expansion) (21/7) | Stage 1A Cohort 01A - Cobimetinib 60 mg (14/14) | Stage 1A Cohort 02A - Cobimetinib 80 mg (14/14) | Stage 1A Cohort 03A - Cobimetinib 100 mg (14/14) | Stage 1A Cohort 04A - Cobimetinib 125 mg (14/14) | Stage 2A Cohort 30 - Cobimetinib 100 mg (Expansion) (14/14) | Stage 3 Cohort 40 - Cobimetinib+Midazolam+Dextromethorphan
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 21 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 21 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Disease Progression | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 16 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Unspecified Reason | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Period: Stage 2A
Arm/Group | Stage 1 Cohort 01 - Cobimetinib 0.05 mg/kg (21/7) | Stage 1 Cohort 02 - Cobimetinib 0.10 mg/kg (21/7) | Stage 1 Cohort 03 - Cobimetinib 0.20 mg/kg (21/7) | Stage 1 Cohort 04 - Cobimetinib 10 mg (21/7) | Stage 1 Cohort 05 - Cobimetinib 20 mg (21/7) | Stage 1 Cohort 06 - Cobimetinib 40 mg (21/7) | Stage 1 Cohort 07 - Cobimetinib 60 mg (21/7) | Stage 1 Cohort 08 - Cobimetinib 80 mg (21/7) | Stage 2 Cohort 20 - Cobimetinib 60 mg (Expansion) (21/7) | Stage 1A Cohort 01A - Cobimetinib 60 mg (14/14) | Stage 1A Cohort 02A - Cobimetinib 80 mg (14/14) | Stage 1A Cohort 03A - Cobimetinib 100 mg (14/14) | Stage 1A Cohort 04A - Cobimetinib 125 mg (14/14) | Stage 2A Cohort 30 - Cobimetinib 100 mg (Expansion) (14/14) | Stage 3 Cohort 40 - Cobimetinib+Midazolam+Dextromethorphan
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 22 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 21 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Disease Progression | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 10 | 0
Not completed — Unspecified Reason | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Period: Stage 3
Arm/Group | Stage 1 Cohort 01 - Cobimetinib 0.05 mg/kg (21/7) | Stage 1 Cohort 02 - Cobimetinib 0.10 mg/kg (21/7) | Stage 1 Cohort 03 - Cobimetinib 0.20 mg/kg (21/7) | Stage 1 Cohort 04 - Cobimetinib 10 mg (21/7) | Stage 1 Cohort 05 - Cobimetinib 20 mg (21/7) | Stage 1 Cohort 06 - Cobimetinib 40 mg (21/7) | Stage 1 Cohort 07 - Cobimetinib 60 mg (21/7) | Stage 1 Cohort 08 - Cobimetinib 80 mg (21/7) | Stage 2 Cohort 20 - Cobimetinib 60 mg (Expansion) (21/7) | Stage 1A Cohort 01A - Cobimetinib 60 mg (14/14) | Stage 1A Cohort 02A - Cobimetinib 80 mg (14/14) | Stage 1A Cohort 03A - Cobimetinib 100 mg (14/14) | Stage 1A Cohort 04A - Cobimetinib 125 mg (14/14) | Stage 2A Cohort 30 - Cobimetinib 100 mg (Expansion) (14/14) | Stage 3 Cohort 40 - Cobimetinib+Midazolam+Dextromethorphan
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 20
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 17
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Disease Progression | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 9
Not completed — Unspecified Reason | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5

BASELINE CHARACTERISTICS:
Population: Safety population consisted of all participants who received at least 1 dose of study drug.
Groups:
- Stage 1 Cohort 01 - Cobimetinib 0.05 mg/kg (21/7): Participants received cobimetinib 0.05 mg/kg via solution or capsule, once daily for Days 1-21 of each 28-day cycle. Treatment was continued until PD or unacceptable toxicity for up to 1 year at the discretion of investigator and beyond 1 year with the agreement of the sponsor.
- Total: Total of all reporting groups
Arm/Group | Stage 1 Cohort 01 - Cobimetinib 0.05 mg/kg (21/7) | Stage 1 Cohort 02 - Cobimetinib 0.10 mg/kg (21/7) | Stage 1 Cohort 03 - Cobimetinib 0.20 mg/kg (21/7) | Stage 1 Cohort 04 - Cobimetinib 10 mg (21/7) | Stage 1 Cohort 05 - Cobimetinib 20 mg (21/7) | Stage 1 Cohort 06 - Cobimetinib 40 mg (21/7) | Stage 1 Cohort 07 - Cobimetinib 60 mg (21/7) | Stage 1 Cohort 08 - Cobimetinib 80 mg (21/7) | Stage 2 Cohort 20 - Cobimetinib 60 mg (Expansion) (21/7) | Stage 1A Cohort 01A - Cobimetinib 60 mg (14/14) | Stage 1A Cohort 02A - Cobimetinib 80 mg (14/14) | Stage 1A Cohort 03A - Cobimetinib 100 mg (14/14) | Stage 1A Cohort 04A - Cobimetinib 125 mg (14/14) | Stage 2A Cohort 30 - Cobimetinib 100 mg (Expansion) (14/14) | Stage 3 Cohort 40 - Cobimetinib+Midazolam+Dextromethorphan | Total
Number analyzed (Participants) | 4 | 3 | 3 | 3 | 3 | 6 | 7 | 7 | 21 | 3 | 3 | 8 | 6 | 22 | 20 | 119
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.0 (11.52) | 60.7 (19.73) | 51.3 (6.35) | 66.0 (10.82) | 60.7 (9.61) | 62.0 (12.38) | 63.9 (5.87) | 54.4 (8.40) | 59.7 (13.08) | 52.7 (13.20) | 49.7 (21.08) | 55.1 (13.46) | 61.5 (13.61) | 61.1 (11.45) | 57.1 (15.60) | 59.1 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 0 | 2 | 3 | 1 | 3 | 2 | 3 | 11 | 1 | 3 | 4 | 4 | 10 | 9 | 59
  Male | 1 | 3 | 1 | 0 | 2 | 3 | 5 | 4 | 10 | 2 | 0 | 4 | 2 | 12 | 11 | 60

OUTCOME MEASURES:

1. Primary Outcome: Stage 1 and 1A: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: Adverse events (AE) were graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) v3.0. DLT was defined as either of the following occurring during the Study Treatment Period. The occurrence of a drug-related AE that, in the opinion of the cohort review committee (CRC), was of potential clinical significance such that further dose escalation would expose participants in higher dose cohorts to risk of irreversible medical harm or require medical treatment to avoid irreversible medical harm or non-hematologic toxicity
  * Grade 3 or 4 events, including Grade 3 nausea and/or vomiting and/or Grade 3 diarrhea, despite prophylaxis and/or treatment Hematologic toxicity
  * Grade 4 thrombocytopenia
  * Grade 4 neutropenia of greater than or equal to (≥) 4 days' duration
  * Grade 4 neutropenia of any duration with fever or documented infection
Time Frame: Stage 1 and 1A: Days 1 to 28 of Cycle 1
Population: Safety population; Stages 1 and 1A participants only.
Measure: Number; unit: participants
Groups:
- Stage 1 Cohort 01 - Cobimetinib 0.05 mg/kg (21/7): Participants received cobimetinib (GDC-0973/XL518) 0.05 mg/kg via solution or capsule, once daily for Days 1-21 of each 28-day cycle (21 days on drug followed by 7 days off treatment [21/7 schedule]). Treatment was continued until progressive disease (PD) or unacceptable toxicity for up to 1 year at the discretion of investigator and beyond 1 year with the agreement of the sponsor.
Arm/Group | Stage 1 Cohort 01 - Cobimetinib 0.05 mg/kg (21/7) | Stage 1 Cohort 02 - Cobimetinib 0.10 mg/kg (21/7) | Stage 1 Cohort 03 - Cobimetinib 0.20 mg/kg (21/7) | Stage 1 Cohort 04 - Cobimetinib 10 mg (21/7) | Stage 1 Cohort 05 - Cobimetinib 20 mg (21/7) | Stage 1 Cohort 06 - Cobimetinib 40 mg (21/7) | Stage 1 Cohort 07 - Cobimetinib 60 mg (21/7) | Stage 1 Cohort 08 - Cobimetinib 80 mg (21/7) | Stage 1A Cohort 01A - Cobimetinib 60 mg (14/14) | Stage 1A Cohort 02A - Cobimetinib 80 mg (14/14) | Stage 1A Cohort 03A - Cobimetinib 100 mg (14/14) | Stage 1A Cohort 04A - Cobimetinib 125 mg (14/14)
Number analyzed (Participants) | 4 | 3 | 3 | 3 | 3 | 6 | 7 | 7 | 3 | 3 | 8 | 6
participants | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 2

2. Primary Outcome: Stage 1: Maximum Tolerated Dose (MTD) of Cobimetinib in 21/7 Schedule
Description: AEs were graded according to the NCI-CTCAE v3.0. A DLT was determined from clinical findings during the Study Treatment Period (Cycle 1, Days 1). MTD was defined as the dose at which no DLTs were observed. DLT was defined as either of the following occurring during the Study Treatment Period. The occurrence of a drug-related AE that, in the opinion of the CRC, was of potential clinical significance such that further dose escalation would expose participants in higher dose cohorts to risk of irreversible medical harm or require medical treatment to avoid irreversible medical harm or non-hematologic toxicity
  * Grade 3 or 4 events, including Grade 3 nausea and/or vomiting and/or Grade 3 diarrhea, despite prophylaxis and/or treatment Hematologic toxicity
  * Grade 4 thrombocytopenia
  * Grade 4 neutropenia of greater than or equal to (≥) 4 days' duration
  * Grade 4 neutropenia of any duration with fever or documented infection
Time Frame: Stage 1: Days 1 to 28 of Cycle 1
Population: Safety population; Stage 1 participants only.
Measure: Number; unit: milligrams (mg)
Groups:
- Stage 1 All Cohorts (21/7): Participants received cobimetinib via solution or capsule, once daily for Days 1-21 of each 28-day cycle and were on 21-days-on and 7-days-off schedule. Treatment was continued until PD or unacceptable toxicity for up to 1 year at the discretion of investigator and beyond 1 year with the agreement of the sponsor.
Arm/Group | Stage 1 All Cohorts (21/7)
Number analyzed (Participants) | 36
milligrams (mg) | 60

3. Primary Outcome: Stage 1A: MTD of Cobimetinib in 14/14 Schedule
Description: AEs were graded according to NCI-CTCAE v3.0. A DLT was the basis for determining MTD in Stage 1A participants. The participants of Stage 1A are dose-escalation cohorts, starting at the MTD of the 21/7 schedule, were treated on a 14/14 schedule to determine the MTD. A DLT was defined as either of the following occurring during the Study Treatment Period:
  Occurrence of a drug-related AE that, in the opinion of the CRC, was of potential clinical significance such that further dose escalation would expose participants to risk of irreversible medical harm; Nonhematologic toxicity: Grade 3 or 4 events, including Grade 3 nausea and/or vomiting and/or Grade 3 diarrhea, despite prophylaxis and/or treatment; Hematologic toxicity: Grade 4 thrombocytopenia. Grade 4 neutropenia of more than 4 days' duration; Grade 4 neutropenia of any duration with fever or documented infection. AEs (Grade 3 or higher) for which a clinical cause unrelated to cobimetinib was evident was not considered DLTs.
Time Frame: Stage 1A: Days 1 to 28 of Cycle 1
Population: Safety population; Stage 1A participants only.
Measure: Number; unit: mg
Groups:
- Stage 1A - All Cohorts (14/14): Participants received cobimetinib via solution or capsule, once daily for Days 1-14 of each 28-day cycle and were on a 14-days-on and 14-days-off schedule. Treatment was continued until PD or unacceptable toxicity for up to 1 year at the discretion of investigator and beyond 1 year with the agreement of the sponsor.
Arm/Group | Stage 1A - All Cohorts (14/14)
Number analyzed (Participants) | 20
mg | 100

4. Primary Outcome: Stage 1: Maximum Observed Concentration (Cmax) of Cobimetinib at Day 1, Cycle 1
Description: Cmax is defined as the maximum plasma concentration achieved after administration of cobimetinib on Day 1, Cycle 1 in Stage 1 and was measured as nanograms per milliliter (ng/mL).
Time Frame: Stage 1: Pre-dose and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12-18 hours post-dose on Cycle 1 Day 1 and pre-dose on Cycle 1 Day 2
Population: Safety population; Stage 1 participants only.
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | Stage 1 Cohort 01 - Cobimetinib 0.05 mg/kg (21/7) | Stage 1 Cohort 02 - Cobimetinib 0.10 mg/kg (21/7) | Stage 1 Cohort 03 - Cobimetinib 0.20 mg/kg (21/7) | Stage 1 Cohort 04 - Cobimetinib 10 mg (21/7) | Stage 1 Cohort 05 - Cobimetinib 20 mg (21/7) | Stage 1 Cohort 06 - Cobimetinib 40 mg (21/7) | Stage 1 Cohort 07 - Cobimetinib 60 mg (21/7) | Stage 1 Cohort 08 - Cobimetinib 80 mg (21/7)
Number analyzed (Participants) | 4 | 3 | 3 | 3 | 3 | 6 | 7 | 7
ng/mL | 4.51 (5.8) | 6.92 (3.8) | 18.3 (13.0) | 18.8 (5.1) | 30.8 (69.0) | 71.7 (57.0) | 163.0 (79.0) | 261.0 (110.0)

5. Primary Outcome: Stage 1: Area Under the Plasma Cobimetinib Concentration Curve From Time 0 to 24 Hours (AUC 0-24) Day 1, Cycle 1
Description: The area under the concentrations-time curve (AUC0-24) was calculated with the measured data points from the time of administration of cobimetinib up to 24 h after administration by the trapezoidal formula. AUC 0-24 is the truncated AUC over a 24-hour sampling interval. The concentration-time curve is the result of time points of blood sampling and its measured concentration of free cobimetinib in the blood samples. AUC is measured as hours times nanograms per milliliter (h*ng/mL).
Time Frame: Stage 1: Pre-dose & 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12-18 hours post-dose on Cycle 1 Day 1, pre-dose on Cycle 1 Day 2
Population: Safety population; Stage 1 participants only.
Measure: Geometric Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Stage 1 Cohort 01 - Cobimetinib 0.05 mg/kg (21/7) | Stage 1 Cohort 02 - Cobimetinib 0.10 mg/kg (21/7) | Stage 1 Cohort 03 - Cobimetinib 0.20 mg/kg (21/7) | Stage 1 Cohort 04 - Cobimetinib 10 mg (21/7) | Stage 1 Cohort 05 - Cobimetinib 20 mg (21/7) | Stage 1 Cohort 06 - Cobimetinib 40 mg (21/7) | Stage 1 Cohort 07 - Cobimetinib 60 mg (21/7) | Stage 1 Cohort 08 - Cobimetinib 80 mg (21/7)
Number analyzed (Participants) | 4 | 3 | 3 | 3 | 3 | 6 | 7 | 7
h*ng/mL | 56.2 (65.0) | 68.0 (47.0) | 203.0 (130.0) | 242.0 (64.0) | 440.0 (870.0) | 785.0 (560.0) | 1620.0 (830.0) | 3060.0 (950.0)

6. Primary Outcome: Stage 1: Time to Maximum Concentration (Tmax) of Cobimetinib at Day 1, Cycle 1
Description: Tmax is defined as the time to reach Cmax during stage 1 at Day 1 Cycle 1.
Time Frame: Stage 1: Pre-dose & 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12-18 hours post-dose on Cycle 1 Day 1 and pre-dose on Cycle 1 Day 2
Population: Safety population; Stage 1 participants only.
Measure: Median (Full Range); unit: hours
Arm/Group | Stage 1 Cohort 01 - Cobimetinib 0.05 mg/kg (21/7) | Stage 1 Cohort 02 - Cobimetinib 0.10 mg/kg (21/7) | Stage 1 Cohort 03 - Cobimetinib 0.20 mg/kg (21/7) | Stage 1 Cohort 04 - Cobimetinib 10 mg (21/7) | Stage 1 Cohort 05 - Cobimetinib 20 mg (21/7) | Stage 1 Cohort 06 - Cobimetinib 40 mg (21/7) | Stage 1 Cohort 07 - Cobimetinib 60 mg (21/7) | Stage 1 Cohort 08 - Cobimetinib 80 mg (21/7)
Number analyzed (Participants) | 4 | 3 | 3 | 3 | 3 | 6 | 7 | 7
hours | 2.0 [2.0 to 8.0] | 1.0 [1.0 to 2.0] | 1.5 [1.0 to 1.5] | 3.0 [1.0 to 4.0] | 4.0 [2.0 to 4.0] | 2.5 [1.5 to 6.0] | 2.0 [1.0 to 4.0] | 2.0 [1.5 to 2.0]

7. Secondary Outcome: Stage 1: Tmax of Cobimetinib at Steady State
Description: Tmax is defined as the time to reach Cmax during stage 1 in steady state. Steady state was reached when overall intake of cobimetinib was in dynamic equilibrium with its elimination.
Time Frame: Stage 1: Pre-dose & 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12-18 hours post-dose on Cycle 1 Day 21, 24, 48, and 72 hours post Cycle 1 Day 21 dose (Cycle 1 Day 22, 23, and 24, respectively)
Population: Safety population; Stage 1 participants only. Number of participants analyzed = participants who were evaluable for this outcome.
Measure: Median (Full Range); unit: hours
Arm/Group | Stage 1 Cohort 01 - Cobimetinib 0.05 mg/kg (21/7) | Stage 1 Cohort 02 - Cobimetinib 0.10 mg/kg (21/7) | Stage 1 Cohort 03 - Cobimetinib 0.20 mg/kg (21/7) | Stage 1 Cohort 04 - Cobimetinib 10 mg (21/7) | Stage 1 Cohort 05 - Cobimetinib 20 mg (21/7) | Stage 1 Cohort 06 - Cobimetinib 40 mg (21/7) | Stage 1 Cohort 07 - Cobimetinib 60 mg (21/7) | Stage 1 Cohort 08 - Cobimetinib 80 mg (21/7)
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 6 | 7 | 7
hours | 4.0 [2.0 to 4.0] | 1.0 [1.0 to 2.0] | 2.25 [1.5 to 3.0] | 4.0 [3.0 to 4.0] | 3.0 [3.0 to 3.0] | 2.0 [1.5 to 3.0] | 3.0 [1.5 to 4.0] | 2.5 [2.0 to 4.0]

8. Secondary Outcome: Stage 1: AUC 0-24 of Cobimetinib at Steady State
Description: The area under the AUC0-24 for steady state in stage 1 was calculated with the measured data points from the time of administration of cobimetinib up to 24 h after administration by the trapezoidal formula. AUC 0-24 is the truncated AUC over a 24-hour sampling interval. The concentration-time curve is the result of time points of blood sampling and its measured concentration of free cobimetinib in the blood samplings.
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Stage 1 Cohort 01 - Cobimetinib 0.05 mg/kg (21/7) | Stage 1 Cohort 02 - Cobimetinib 0.10 mg/kg (21/7) | Stage 1 Cohort 03 - Cobimetinib 0.20 mg/kg (21/7) | Stage 1 Cohort 04 - Cobimetinib 10 mg (21/7) | Stage 1 Cohort 05 - Cobimetinib 20 mg (21/7) | Stage 1 Cohort 06 - Cobimetinib 40 mg (21/7) | Stage 1 Cohort 07 - Cobimetinib 60 mg (21/7) | Stage 1 Cohort 08 - Cobimetinib 80 mg (21/7)
Number analyzed (Participants) | 3 | 3 | 2 | 3 | 1 | 5 | 4 | 6
h*ng/mL | 202.0 (158.0) | 288.0 (200.0) | 411.0 (199.0) | 763.0 (168.0) | 886.0 | 5370.0 (4600.0) | 6250.0 (3540.0) | 10500.0 (10500.0)

9. Secondary Outcome: Stage 1: AUC 0-24/D of Cobimetinib at Steady State
Description: AUC 0-24/D is the dose normalized truncated AUC over a 24-hour sampling interval.
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: ng*hr/mL/mg
Arm/Group | Stage 1 Cohort 01 - Cobimetinib 0.05 mg/kg (21/7) | Stage 1 Cohort 02 - Cobimetinib 0.10 mg/kg (21/7) | Stage 1 Cohort 03 - Cobimetinib 0.20 mg/kg (21/7) | Stage 1 Cohort 04 - Cobimetinib 10 mg (21/7) | Stage 1 Cohort 05 - Cobimetinib 20 mg (21/7) | Stage 1 Cohort 06 - Cobimetinib 40 mg (21/7) | Stage 1 Cohort 07 - Cobimetinib 60 mg (21/7) | Stage 1 Cohort 08 - Cobimetinib 80 mg (21/7)
Number analyzed (Participants) | 3 | 3 | 2 | 3 | 1 | 5 | 4 | 6
ng*hr/mL/mg | 62.4 (36.3) | 34 (16.9) | 28.2 (8.43) | 76.3 (16.8) | 44.3 | 134 (115) | 104 (59.1) | 132 (131)

10. Secondary Outcome: Stage 1: Accumulation Ratio of Cobimetinib at Steady State
Description: Accumulation Ratio: AUC0-24 at steady state divided by AUC0-24 on Cycle 1 Day 1. It was calculated only for participants who had a quantifiable AUC 0-24 at steady state.
Time Frame: Stage 1: Pre-dose & 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12-18 hours post-dose on Cycle 1 Day 1, Day 21, 24, 48, and 72 hours post Cycle 1 Day 21 dose (Cycle 1 Day 22, 23, and 24, respectively)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Stage 1 Cohort 01 - Cobimetinib 0.05 mg/kg (21/7) | Stage 1 Cohort 02 - Cobimetinib 0.10 mg/kg (21/7) | Stage 1 Cohort 03 - Cobimetinib 0.20 mg/kg (21/7) | Stage 1 Cohort 04 - Cobimetinib 10 mg (21/7) | Stage 1 Cohort 05 - Cobimetinib 20 mg (21/7) | Stage 1 Cohort 06 - Cobimetinib 40 mg (21/7) | Stage 1 Cohort 07 - Cobimetinib 60 mg (21/7) | Stage 1 Cohort 08 - Cobimetinib 80 mg (21/7)
Number analyzed (Participants) | 3 | 3 | 2 | 3 | 1 | 4 | 4 | 5
ratio | 3.56 (1.76) | 3.66 (0.901) | 2.65 (0.886) | 3.23 (1.03) | 2.96 | 3.61 (2.27) | 2.87 (0.787) | 3.26 (2.1)

11. Secondary Outcome: Stage 1: Apparent Clearance of Cobimetinib at Steady State
Description: Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood. Apparent clearance was calculated only for participants who had a quantifiable AUC 0-24 in steady state.
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Liters per hour (L/hr)
Arm/Group | Stage 1 Cohort 01 - Cobimetinib 0.05 mg/kg (21/7) | Stage 1 Cohort 02 - Cobimetinib 0.10 mg/kg (21/7) | Stage 1 Cohort 03 - Cobimetinib 0.20 mg/kg (21/7) | Stage 1 Cohort 04 - Cobimetinib 10 mg (21/7) | Stage 1 Cohort 05 - Cobimetinib 20 mg (21/7) | Stage 1 Cohort 06 - Cobimetinib 40 mg (21/7) | Stage 1 Cohort 07 - Cobimetinib 60 mg (21/7) | Stage 1 Cohort 08 - Cobimetinib 80 mg (21/7)
Number analyzed (Participants) | 3 | 3 | 2 | 3 | 1 | 5 | 4 | 6
Liters per hour (L/hr) | 22.4 (17.2) | 34.0 (14.2) | 37.1 (11.1) | 13.5 (2.71) | 22.6 | 14.0 (10.1) | 11.8 (5.71) | 11.6 (5.42)

12. Secondary Outcome: Stage 1: Half-Life (t1/2) of Cobimetinib at Steady State
Description: t1/2 is the half-life of cobimetinib measured over the terminal phase by noncompartmental analysis in stage 1 in steady state.
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Median (Full Range); unit: hours
Arm/Group | Stage 1 Cohort 01 - Cobimetinib 0.05 mg/kg (21/7) | Stage 1 Cohort 02 - Cobimetinib 0.10 mg/kg (21/7) | Stage 1 Cohort 03 - Cobimetinib 0.20 mg/kg (21/7) | Stage 1 Cohort 04 - Cobimetinib 10 mg (21/7) | Stage 1 Cohort 05 - Cobimetinib 20 mg (21/7) | Stage 1 Cohort 06 - Cobimetinib 40 mg (21/7) | Stage 1 Cohort 07 - Cobimetinib 60 mg (21/7) | Stage 1 Cohort 08 - Cobimetinib 80 mg (21/7)
Number analyzed (Participants) | 1 | 3 | 2 | 3 | 1 | 5 | 4 | 5
hours | 80.0 [80.0 to 80.0] | 64.0 [51.5 to 73] | 47.8 [46.5 to 49.1] | 66.0 [34.0 to 67.5] | 50.5 [50.5 to 50.5] | 41.3 [34.2 to 62.4] | 51.3 [23.1 to 61.4] | 60.0 [33.5 to 65.4]

13. Secondary Outcome: Stage 1: Cmax of Cobimetinib at Steady State
Description: Cmax is defined as the maximum plasma concentration achieved after administration of cobimetinib in Stage 1 and was measured at steady state in ng/mL.
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Stage 1 Cohort 01 - Cobimetinib 0.05 mg/kg (21/7) | Stage 1 Cohort 02 - Cobimetinib 0.10 mg/kg (21/7) | Stage 1 Cohort 03 - Cobimetinib 0.20 mg/kg (21/7) | Stage 1 Cohort 04 - Cobimetinib 10 mg (21/7) | Stage 1 Cohort 05 - Cobimetinib 20 mg (21/7) | Stage 1 Cohort 06 - Cobimetinib 40 mg (21/7) | Stage 1 Cohort 07 - Cobimetinib 60 mg (21/7) | Stage 1 Cohort 08 - Cobimetinib 80 mg (21/7)
Number analyzed (Participants) | 3 | 3 | 2 | 3 | 1 | 5 | 4 | 6
ng/mL | 13.5 (9.53) | 19.8 (15.2) | 28.7 (8.63) | 53.0 (5.4) | 54.7 | 341.0 (244.0) | 401.0 (214.0) | 641.0 (514.0)

14. Secondary Outcome: Stage 1A: Tmax of Cobimetinib at Cycle 1 Day 1
Description: Tmax is defined as the time to reach Cmax during stage 1A at Day 1.
Time Frame: Stage 1A: Pre-dose & 0.5, 1, 1.5, 2, 3, 4, 6 hours post-dose on Cycle 1 Day 1, pre-dose on Cycle 1 Day 2
Population: Safety population; Stage 1A participants only.
Measure: Median (Full Range); unit: hours
Arm/Group | Stage 1A Cohort 01A - Cobimetinib 60 mg (14/14) | Stage 1A Cohort 02A - Cobimetinib 80 mg (14/14) | Stage 1A Cohort 03A - Cobimetinib 100 mg (14/14) | Stage 1A Cohort 04A - Cobimetinib 125 mg (14/14)
Number analyzed (Participants) | 3 | 3 | 8 | 6
hours | 3.0 [1.5 to 4.0] | 4.0 [2.0 to 24] | 3.5 [1.5 to 6] | 2.5 [2.0 to 4.0]

15. Secondary Outcome: Stage 1A: Cmax of Cobimetinib at Cycle 1 Day 1
Description: Cmax is defined as the maximum plasma concentration achieved after administration of cobimetinib on on Day 1 in Stage 1A and was measured as ng/mL.
Time Frame: Stage 1A: Pre-dose & 0.5, 1, 1.5, 2, 3, 4, 6 hours post-dose on Cycle 1 Day 1, pre-dose on Cycle 1 Day 2
Population: Safety population; Stage 1A participants only.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Stage 1A Cohort 01A - Cobimetinib 60 mg (14/14) | Stage 1A Cohort 02A - Cobimetinib 80 mg (14/14) | Stage 1A Cohort 03A - Cobimetinib 100 mg (14/14) | Stage 1A Cohort 04A - Cobimetinib 125 mg (14/14)
Number analyzed (Participants) | 3 | 3 | 8 | 6
ng/mL | 78.4 (88.0) | 167.0 (63.0) | 258.0 (140.0) | 533.0 (347.0)

16. Secondary Outcome: Stage 1A: AUC 0-24 of Cobimetinib at Cycle 1 Day 1
Description: AUC0-24 for stage 1A was calculated on Day 1 with the measured data points from the time of administration of cobimetinib up to 24 h after administration by the trapezoidal formula. AUC 0-24 is the truncated AUC over a 24-hour sampling interval. The concentration-time curve is the result of time points of blood sampling and its measured concentration of free cobimetinib in the blood samplings.
Time Frame: Stage 1A: Pre-dose & 0.5, 1, 1.5, 2, 3, 4, 6 hours post-dose on Cycle 1 Day 1, pre-dose on Cycle 1 Day 2
Population: Safety population; Stage 1A participants only.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Stage 1A Cohort 01A - Cobimetinib 60 mg (14/14) | Stage 1A Cohort 02A - Cobimetinib 80 mg (14/14) | Stage 1A Cohort 03A - Cobimetinib 100 mg (14/14) | Stage 1A Cohort 04A - Cobimetinib 125 mg (14/14)
Number analyzed (Participants) | 3 | 3 | 8 | 6
h*ng/mL | 1140 (1150) | 2130 (70.1) | 4020 (2000) | 7190 (3640)

17. Secondary Outcome: Stage 1A: t1/2 of Cobimetinib at Steady State
Description: t1/2 is the half-life of cobimetinib measured over the terminal phase by noncompartmental analysis in stage 1A in steady state.
Time Frame: Stage 1A: Pre-dose & 0.5, 1, 1.5, 2, 3, 4, 6 hours post-dose on Cycle 1 Day 14, 24, 48, 72 hours post Cycle 1 Day 14 dose (Cycle 1 Day 15, 16, and 17, respectively)
Population: Safety population; Stage 1A participants only. Number of participants analyzed = participants who were evaluable for this outcome.
Measure: Median (Full Range); unit: hours
Arm/Group | Stage 1A Cohort 01A - Cobimetinib 60 mg (14/14) | Stage 1A Cohort 02A - Cobimetinib 80 mg (14/14) | Stage 1A Cohort 03A - Cobimetinib 100 mg (14/14) | Stage 1A Cohort 04A - Cobimetinib 125 mg (14/14)
Number analyzed (Participants) | 1 | 1 | 3 | 1
hours | 59.4 [59.4 to 59.4] | 44.1 [44.1 to 44.1] | 51.6 [48.1 to 71.1] | 47.7 [47.7 to 47.7]

18. Secondary Outcome: Stage 1A: Tmax of Cobimetinib at Steady State
Description: Tmax is defined as the time to reach Cmax during stage 1A in steady state.
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Median (Full Range); unit: hours
Arm/Group | Stage 1A Cohort 01A - Cobimetinib 60 mg (14/14) | Stage 1A Cohort 02A - Cobimetinib 80 mg (14/14) | Stage 1A Cohort 03A - Cobimetinib 100 mg (14/14) | Stage 1A Cohort 04A - Cobimetinib 125 mg (14/14)
Number analyzed (Participants) | 3 | 3 | 5 | 3
hours | 2.0 [1.5 to 4.0] | 2.0 [2.0 to 6.0] | 3 [1.5 to 4.0] | 6 [2.0 to 6.0]

19. Secondary Outcome: Stage 1A: Apparent Clearance of Cobimetinib at Steady State
Description: as for outcome 11
Time Frame: as for outcome 17
Population: Safety population; Stage 1A participants only. Number pf participants analyzed = participants who were evaluable for this outcome.
Measure: Mean (Standard Deviation); unit: L/hr
Arm/Group | Stage 1A Cohort 01A - Cobimetinib 60 mg (14/14) | Stage 1A Cohort 02A - Cobimetinib 80 mg (14/14) | Stage 1A Cohort 03A - Cobimetinib 100 mg (14/14) | Stage 1A Cohort 04A - Cobimetinib 125 mg (14/14)
Number analyzed (Participants) | 3 | 3 | 5 | 3
L/hr | 25.1 (13.5) | 14.9 (8.33) | 21.9 (20.3) | 6.9 (3.22)

20. Secondary Outcome: Stage 1A: Accumulation Ratio of Cobimetinib at Steady State
Description: as for outcome 10
Time Frame: Stage 1A: Pre-dose & 0.5, 1, 1.5, 2, 3, 4, 6 hours post-dose on Cycle 1 Day 1, 14, 24, 48, 72 hours post Cycle 1 Day 14 dose (Cycle 1 Day 15, 16, and 17, respectively)
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Stage 1A Cohort 01A - Cobimetinib 60 mg (14/14) | Stage 1A Cohort 02A - Cobimetinib 80 mg (14/14) | Stage 1A Cohort 03A - Cobimetinib 100 mg (14/14) | Stage 1A Cohort 04A - Cobimetinib 125 mg (14/14)
Number analyzed (Participants) | 3 | 3 | 5 | 3
ratio | 2.32 (0.448) | 3.14 (1.77) | 2.6 (2.32) | 5.15 (2.08)

21. Secondary Outcome: Stage 1A: AUC 0-24 of Cobimetinib at Steady State
Description: The area under the AUC0-24 for steady state in stage 1A was calculated with the measured data points from the time of administration of cobimetinib up to 24 h after administration by the trapezoidal formula. AUC 0-24 is the truncated AUC over a 24-hour sampling interval. The concentration-time curve is the result of time points of blood sampling and its measured concentration of free cobimetinib in the blood samplings.
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Stage 1A Cohort 01A - Cobimetinib 60 mg (14/14) | Stage 1A Cohort 02A - Cobimetinib 80 mg (14/14) | Stage 1A Cohort 03A - Cobimetinib 100 mg (14/14) | Stage 1A Cohort 04A - Cobimetinib 125 mg (14/14)
Number analyzed (Participants) | 3 | 3 | 5 | 3
h*ng/mL | 2990.0 (1750.0) | 6740.0 (3830.0) | 11500.0 (10500.0) | 21500.0 (11300.0)

22. Secondary Outcome: Stage 1A: AUC 0-24/D of Cobimetinib at Steady State
Description: AUC 0-24/D is the dose normalized truncated AUC over a 24-hour sampling interval.
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: ng*hr/mL/mg
Arm/Group | Stage 1A Cohort 01A - Cobimetinib 60 mg (14/14) | Stage 1A Cohort 02A - Cobimetinib 80 mg (14/14) | Stage 1A Cohort 03A - Cobimetinib 100 mg (14/14) | Stage 1A Cohort 04A - Cobimetinib 125 mg (14/14)
Number analyzed (Participants) | 3 | 3 | 5 | 3
ng*hr/mL/mg | 49.8 (29.2) | 84.2 (47.8) | 115.0 (105.0) | 172.0 (90.4)

23. Secondary Outcome: Stage 1A: Cmax of Cobimetinib at Steady State
Description: Cmax is defined as the maximum plasma concentration achieved after administration of cobimetinib in Stage 1A and was measured in steady state as ng/mL.
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Stage 1A Cohort 01A - Cobimetinib 60 mg (14/14) | Stage 1A Cohort 02A - Cobimetinib 80 mg (14/14) | Stage 1A Cohort 03A - Cobimetinib 100 mg (14/14) | Stage 1A Cohort 04A - Cobimetinib 125 mg (14/14)
Number analyzed (Participants) | 3 | 3 | 5 | 3
ng/mL | 180.0 (101.0) | 494.0 (175.0) | 640.0 (511.0) | 1160.0 (540.0)

24. Secondary Outcome: Stage 2: Cmax of Cobimetinib at Cycle 1 Day 1
Description: Cmax is defined as the maximum plasma concentration achieved after administration of cobimetinib in Stage 2 and was measured in ng/mL.
Time Frame: Stage 2: Pre-dose & 0.5, 1, 1.5, 2, 3, 4, 6 hours post-dose on Cycle 1 Day 1, pre-dose on Cycle 1 Day 2
Population: Safety population; Stage 2 participants only. Number of participants analyzed = participants who were evaluable for this outcome.
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | Stage 2 Cohort 20 - Cobimetinib 60 mg (Expansion) (21/7)
Number analyzed (Participants) | 19
ng/mL | 184.0 (160.0)

25. Secondary Outcome: Stage 2:AUC 0-24 of Cobimetinib at Cycle 1 Day 1
Description: The area under the AUC0-24 on Day 1 in stage 2 was calculated with the measured data points from the time of administration of cobimetinib up to 24 h after administration by the trapezoidal formula. AUC 0-24 is the truncated AUC over a 24-hour sampling interval. The concentration-time curve is the result of time points of blood sampling and its measured concentration of free cobimetinib in the blood samplings.
Time Frame: Stage 2: Pre-dose & 0.5, 1, 1.5, 2, 3, 4, 6 hours post-dose on Cycle 1 Day 1, pre-dose on Cycle 1 Day 2
Population: as for outcome 24
Measure: Geometric Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Stage 2 Cohort 20 - Cobimetinib 60 mg (Expansion) (21/7)
Number analyzed (Participants) | 19
h*ng/mL | 3060.0 (2110.0)

26. Secondary Outcome: Stage 2: Tmax of Cobimetinib at Cycle 1 Day 1
Description: Tmax is defined as the time to reach Cmax during stage 2 on Day 1.
Time Frame: Stage 2: Pre-dose & 0.5, 1, 1.5, 2, 3, 4, 6 hours post-dose on Cycle 1 Day 1, pre-dose on Cycle 1 Day 2
Population: as for outcome 24
Measure: Median (Full Range); unit: hours
Arm/Group | Stage 2 Cohort 20 - Cobimetinib 60 mg (Expansion) (21/7)
Number analyzed (Participants) | 19
hours | 3.0 [1.0 to 6.0]

27. Secondary Outcome: Stage 2: Tmax of Cobimetinib at Steady State
Description: Tmax is defined as the time to reach Cmax during stage 2 in steady state.
Time Frame: Stage 2: Pre-dose & 0.5, 1, 1.5, 2, 3, 4, 6 hours post-dose on Cycle 1 Day 21, 24 hours post Cycle 1 Day 21 dose (Cycle 1 Day 22), and between Cycle 1 Days 26-28
Population: Safety population; Stage 2 participants only; Number of participants analyzed = participants who were evaluable for this outcome.
Measure: Median (Full Range); unit: hours
Arm/Group | Stage 2 Cohort 20 - Cobimetinib 60 mg (Expansion) (21/7)
Number analyzed (Participants) | 13
hours | 4.0 [1.5 to 6.0]

28. Secondary Outcome: Stage 2: AUC 0-24 of Cobimetinib at Steady State
Description: The area under the AUC0-24 for steady state in stage 2 was calculated with the measured data points from the time of administration of cobimetinib up to 24 h after administration by the trapezoidal formula. AUC 0-24 is the truncated AUC over a 24-hour sampling interval. The concentration-time curve is the result of time points of blood sampling and its measured concentration of free cobimetinib in the blood samplings.
Time Frame: as for outcome 27
Population: as for outcome 24
Measure: Geometric Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Stage 2 Cohort 20 - Cobimetinib 60 mg (Expansion) (21/7)
Number analyzed (Participants) | 13
h*ng/mL | 10200.0 (5630.0)

29. Secondary Outcome: Stage 2: AUC 0-24/D of Cobimetinib at Steady State
Description: AUC 0-24/D is the dose normalized truncated AUC over a 24-hour sampling interval.
Time Frame: as for outcome 27
Population: as for outcome 24
Measure: Geometric Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Stage 2 Cohort 20 - Cobimetinib 60 mg (Expansion) (21/7)
Number analyzed (Participants) | 13
h*ng/mL | 102.0 (56.3)

30. Secondary Outcome: Stage 2: Accumulation Ratio of Cobimetinib at Steady State
Description: Accumulation ratio is AUC0-24 at steady state divided by AUC0-24 on Cycle 1 Day 1. It was calculated only for participants who had a quantifiable AUC 0-24 at steady state.
Time Frame: as for outcome 27
Population: as for outcome 24
Measure: Geometric Mean (Standard Deviation); unit: ratio
Arm/Group | Stage 2 Cohort 20 - Cobimetinib 60 mg (Expansion) (21/7)
Number analyzed (Participants) | 13
ratio | 2.5 (0.9)

31. Secondary Outcome: Stage 2: Apparent Clearance of Cobimetinib at Steady State
Description: as for outcome 11
Time Frame: as for outcome 27
Population: Safety population
Measure: Mean (Standard Deviation); unit: L/hr
Arm/Group | Stage 2 Cohort 20 - Cobimetinib 60 mg (Expansion) (21/7)
Number analyzed (Participants) | 13
L/hr | 9.8 (9.9)

32. Secondary Outcome: Stage 2:Half-Life of Cobimetinib at Steady State
Description: T1/2 half-life of cobimetinib measured over the terminal phase by noncompartmental analysis.
Time Frame: as for outcome 27
Population: as for outcome 24
Measure: Median (Full Range); unit: hours
Arm/Group | Stage 2 Cohort 20 - Cobimetinib 60 mg (Expansion) (21/7)
Number analyzed (Participants) | 13
hours | 53.4 [45.3 to 68.3]

33. Secondary Outcome: Stage 2A: AUC 0-24/D of Cobimetinib at Steady State
Description: AUC 0-24/D is the dose normalized truncated AUC over a 24-hour sampling interval.
Time Frame: Stage 2A: Pre-dose & 0.5, 1, 1.5, 2, 3, 4, 6 hours post-dose on Cycle 1 Day 14, 24 hours post Cycle 1 Day 14 dose (Cycle 1 Day 15), and between Cycle 1 Days 26-28
Population: Safety population; Stage 2A participants only. Number of participants analyzed = participants who were evaluable for this outcome.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Stage 2A Cohort 30 - Cobimetinib 100 mg (Expansion) (14/14)
Number analyzed (Participants) | 15
h*ng/mL | 84.8 (52.0)

34. Secondary Outcome: Stage 2A: Accumulation Ratio of Cobimetinib at Steady State
Description: Accumulation Ratio AUC0-24 is ratio of AUC on Day 20: Day 1.
Time Frame: as for outcome 33
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Stage 2A Cohort 30 - Cobimetinib 100 mg (Expansion) (14/14)
Number analyzed (Participants) | 15
ratio | 2.3 (1.2)

35. Secondary Outcome: Stage 2A: Apparent Clearance of Cobimetinib at Steady State
Description: Apparent clearance is the plasma clearance of absorbed drug.
Time Frame: as for outcome 33
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: L/hr
Arm/Group | Stage 2A Cohort 30 - Cobimetinib 100 mg (Expansion) (14/14)
Number analyzed (Participants) | 15
L/hr | 11.8 (5.2)

36. Secondary Outcome: Stage 2A: Half-Life of Cobimetinib at Steady State
Time Frame: as for outcome 33
Population: as for outcome 33
Measure: Median (Full Range); unit: hours
Arm/Group | Stage 2A Cohort 30 - Cobimetinib 100 mg (Expansion) (14/14)
Number analyzed (Participants) | 15
hours | 42.7 [27.8 to 69.6]

37. Secondary Outcome: Stage 2A: Tmax of Cobimetinib at Steady State
Description: Tmax is defined as the time to reach Cmax during stage 2A in steady state.
Time Frame: as for outcome 33
Population: as for outcome 33
Measure: Median (Full Range); unit: hours
Arm/Group | Stage 2A Cohort 30 - Cobimetinib 100 mg (Expansion) (14/14)
Number analyzed (Participants) | 15
hours | 3.0 [1.0 to 6.0]

38. Secondary Outcome: Stage 2A: Cmax of Cobimetinib at Steady State
Description: Cmax is the maximum plasma concentration achieved following the Day 20 dose in Stage 2A.
Time Frame: as for outcome 33
Population: Analysis population; Stage 2A participants only. Number of participants analyzed = participants who were evaluable for this outcome.
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | Stage 2A Cohort 30 - Cobimetinib 100 mg (Expansion) (14/14)
Number analyzed (Participants) | 15
ng/mL | 315.0 (220.0)

39. Secondary Outcome: Stage III: Cmax of Dextromethorphan
Description: Cmax is defined as maximum observed plasma concentration and was determined both in the presence (Cycle 1 Day 15) and absence of cobimetinib (Cycle 1 Day 1).
Time Frame: Stage III: Predose, 0.5, 1, 1.5, 2, 4, 6, 8, and 24 hours after dextromethorphan administration on Days 1 and 15 of Cycle 1
Population: Safety population; Stage 3 participants only. n=number of participants analyzed for specified category.
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | Stage 3 Cohort 40 - Cobimetinib+Midazolam+Dextromethorphan
Number analyzed (Participants) | 20
ng/mL
  With cobimetinib - Cycle 1 Day 15(n=17) | 3.44 (150.0)
  Without cobimetinib - Cycle 1 Day 1 (n=20) | 3.16 (273.0)

40. Secondary Outcome: Stage III: AUC 0-24 of Dextromethorphan
Description: AUC0-24 is the area under the plasma drug concentration curve over a 24-hour sampling interval and was determined both in presence (Cycle 1 Day 15) and absence (Cycle 1 Day 1) of cobimetinib.
Time Frame: as for outcome 39
Population: Safety population; Stage 3 participants only. n = number of participants analyzed for specified category. Number of participants analyzed = participants who were evaluable for this outcome.
Measure: Geometric Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Stage 3 Cohort 40 - Cobimetinib+Midazolam+Dextromethorphan
Number analyzed (Participants) | 19
h*ng/mL
  With cobimetinib - Cycle 1 Day 1 (n=17) | 24.8 (180.0)
  Without cobimetinib - Cycle 1 Day1 (n=19) | 25.8 (240)

41. Secondary Outcome: Stage III: AUC 0-inf of Dextromethorphan
Description: AUC0-inf is AUC from time 0 to infinity and was calculated both in presence Cycle 1 Day 15) and absence (Cycle 1 Day 1) of cobimetinib.
Time Frame: as for outcome 39
Population: as for outcome 40
Measure: Geometric Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Stage 3 Cohort 40 - Cobimetinib+Midazolam+Dextromethorphan
Number analyzed (Participants) | 19
h*ng/mL
  With cobimetinib - Cycle 1 Day 15 (n=13) | 29.1 (250.0)
  Without cobimetinib - Cycle 1 Day1 (n=19) | 18.9 (124.0)

42. Secondary Outcome: Stage III: Cmax of Midazolam
Description: Cmax is the maximum observed plasma concentration and was calculated both in the presence (Cycle 1 Day 15) and absence (Cycle 1 Day 1) of cobimetinib.
Time Frame: as for outcome 39
Population: as for outcome 40
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | Stage 3 Cohort 40 - Cobimetinib+Midazolam+Dextromethorphan
Number analyzed (Participants) | 20
ng/mL
  With cobimetinib - Cycle 1 Day15 (n=17) | 11.5 (64.0)
  Without cobimetinib - Cycle 1 Day 1(n=20) | 10.9 (79.0)

43. Secondary Outcome: Stage III: AUC0-24 of Midazolam
Description: AUC0-24 is the area under the plasma drug concentration curve over a 24-hour sampling interval and was calculated both in the presence (Cycle 1 Day 15) and absence (CXycle 1 Day 1) of cobimetinib.
Time Frame: as for outcome 39
Population: as for outcome 40
Measure: Geometric Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Stage 3 Cohort 40 - Cobimetinib+Midazolam+Dextromethorphan
Number analyzed (Participants) | 14
h*ng/mL
  With cobimetinib - Cycle 1 Day 15 (n=14) | 33.0 (74.0)
  Without cobimetinib - Cycle 1 Day 1 (n=11) | 33.4 (88.0)

44. Secondary Outcome: Stage III: AUC0-inf of Midazolam
Description: AUC0-inf is the AUC from time 0 to infinity and was calculated both in the presence (Cycle 1 Day 15) and absence (Cycle 1 Day 1) of cobimetinib.
Time Frame: as for outcome 39
Population: as for outcome 40
Measure: Geometric Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Stage 3 Cohort 40 - Cobimetinib+Midazolam+Dextromethorphan
Number analyzed (Participants) | 19
h*ng/mL
  With cobimetinib - Cycle 1 Day 15 (n=17) | 34.9 (77.0)
  Without cobimetinib Cycle 1 Day 1 (n=19) | 35.7 (91.0)

ADVERSE EVENTS:
Time Frame: AEs were recorded from the Day 1 of treatment period until the 30 plus or minus 4 days after the last treatment (up to approximately 6 years) .
Groups:
- Stage 3 Cohort 40 - Cobimetinib+Midazolam+Dextromethorphan: Participants received a single dose of midazolam (2 mg of midazolam syrup) and dextromethorphan (30 mg tablet) on Cycle 1 Day 1, in the absence of cobimetinib. After a 2-day washout period, participants received 21 consecutive daily doses of cobimetinib (60-mg) followed by a 7-day washout period. Participants received another single dose of midazolam and dextromethorphan on Cycle 1 Day 15, in the presence of steady-state cobimetinib concentrations. in Cycle 2 and beyond received cobimetinib alone, administered as a 60-mg daily dose for 21 consecutive days in 28-day cycles.
Arm/Group | Stage 1 Cohort 01 - Cobimetinib 0.05 mg/kg (21/7) | Stage 1 Cohort 02 - Cobimetinib 0.10 mg/kg (21/7) | Stage 1 Cohort 03 - Cobimetinib 0.20 mg/kg (21/7) | Stage 1 Cohort 04 - Cobimetinib 10 mg (21/7) | Stage 1 Cohort 05 - Cobimetinib 20 mg (21/7) | Stage 1 Cohort 06 - Cobimetinib 40 mg (21/7) | Stage 1 Cohort 07 - Cobimetinib 60 mg (21/7) | Stage 1 Cohort 08 - Cobimetinib 80 mg (21/7) | Stage 2 Cohort 20 - Cobimetinib 60 mg (Expansion) (21/7) | Stage 1A Cohort 01A - Cobimetinib 60 mg (14/14) | Stage 1A Cohort 02A - Cobimetinib 80 mg (14/14) | Stage 1A Cohort 03A - Cobimetinib 100 mg (14/14) | Stage 1A Cohort 04A - Cobimetinib 125 mg (14/14) | Stage 2A Cohort 30 - Cobimetinib 100 mg (Expansion) (14/14) | Stage 3 Cohort 40 - Cobimetinib+Midazolam+Dextromethorphan
Serious Adverse Events (participants affected / at risk) | 2/4 | 0/3 | 1/3 | 0/3 | 1/3 | 3/6 | 3/7 | 5/7 | 7/21 | 0/3 | 1/3 | 4/8 | 3/6 | 11/22 | 8/20
Other Adverse Events (participants affected / at risk) | 4/4 | 3/3 | 3/3 | 3/3 | 3/3 | 6/6 | 7/7 | 7/7 | 20/21 | 3/3 | 3/3 | 8/8 | 6/6 | 21/22 | 18/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stage 1 Cohort 01 - Cobimetinib 0.05 mg/kg (21/7) (N=4) | Stage 1 Cohort 02 - Cobimetinib 0.10 mg/kg (21/7) (N=3) | Stage 1 Cohort 03 - Cobimetinib 0.20 mg/kg (21/7) (N=3) | Stage 1 Cohort 04 - Cobimetinib 10 mg (21/7) (N=3) | Stage 1 Cohort 05 - Cobimetinib 20 mg (21/7) (N=3) | Stage 1 Cohort 06 - Cobimetinib 40 mg (21/7) (N=6) | Stage 1 Cohort 07 - Cobimetinib 60 mg (21/7) (N=7) | Stage 1 Cohort 08 - Cobimetinib 80 mg (21/7) (N=7) | Stage 2 Cohort 20 - Cobimetinib 60 mg (Expansion) (21/7) (N=21) | Stage 1A Cohort 01A - Cobimetinib 60 mg (14/14) (N=3) | Stage 1A Cohort 02A - Cobimetinib 80 mg (14/14) (N=3) | Stage 1A Cohort 03A - Cobimetinib 100 mg (14/14) (N=8) | Stage 1A Cohort 04A - Cobimetinib 125 mg (14/14) (N=6) | Stage 2A Cohort 30 - Cobimetinib 100 mg (Expansion) (14/14) (N=22) | Stage 3 Cohort 40 - Cobimetinib+Midazolam+Dextromethorphan (N=20)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Faecal incontinence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Generalised oedema (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bile duct obstruction (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Feeding tube complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Troponin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hepatic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pleurodesis (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Peripheral artery thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Stage 1 Cohort 01 - Cobimetinib 0.05 mg/kg (21/7) (N=4) | Stage 1 Cohort 02 - Cobimetinib 0.10 mg/kg (21/7) (N=3) | Stage 1 Cohort 03 - Cobimetinib 0.20 mg/kg (21/7) (N=3) | Stage 1 Cohort 04 - Cobimetinib 10 mg (21/7) (N=3) | Stage 1 Cohort 05 - Cobimetinib 20 mg (21/7) (N=3) | Stage 1 Cohort 06 - Cobimetinib 40 mg (21/7) (N=6) | Stage 1 Cohort 07 - Cobimetinib 60 mg (21/7) (N=7) | Stage 1 Cohort 08 - Cobimetinib 80 mg (21/7) (N=7) | Stage 2 Cohort 20 - Cobimetinib 60 mg (Expansion) (21/7) (N=21) | Stage 1A Cohort 01A - Cobimetinib 60 mg (14/14) (N=3) | Stage 1A Cohort 02A - Cobimetinib 80 mg (14/14) (N=3) | Stage 1A Cohort 03A - Cobimetinib 100 mg (14/14) (N=8) | Stage 1A Cohort 04A - Cobimetinib 125 mg (14/14) (N=6) | Stage 2A Cohort 30 - Cobimetinib 100 mg (Expansion) (14/14) (N=22) | Stage 3 Cohort 40 - Cobimetinib+Midazolam+Dextromethorphan (N=20)
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 1 | 2 | 2 | 3 | 4 | 4 | 13 | 1 | 1 | 6 | 6 | 17 | 12
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 2 | 0 | 1 | 3 | 3 | 7 | 0 | 2 | 6 | 1 | 9 | 4
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 1 | 2 | 3 | 1 | 5 | 0 | 2 | 4 | 2 | 12 | 5
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 2 | 2 | 0 | 0 | 5 | 1 | 9 | 3
Constipation (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 1 | 1 | 3 | 0 | 3 | 0 | 1 | 2 | 0 | 6 | 4
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 3 | 0 | 1 | 2 | 1 | 2 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 4
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 1
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1
Retching (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Anorectal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Faecal incontinence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tongue disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 0 | 0 | 3 | 5 | 5 | 13 | 2 | 2 | 4 | 3 | 11 | 6
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 2 | 0 | 1 | 2 | 3 | 1 | 1 | 0 | 1 | 1 | 2 | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 2 | 3 | 5
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 1 | 1 | 1 | 1 | 3
Skin fissures (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Facial wasting (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nail discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Papule (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Yellow skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 2 | 2 | 0 | 2 | 1 | 2 | 4 | 3 | 10 | 0 | 2 | 6 | 2 | 14 | 8
Oedema peripheral (General disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 4 | 5 | 6 | 1 | 0 | 5 | 1 | 5 | 4
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 3 | 2
Oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 3 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 2
Chills (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 0
Face oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 1
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Feeling hot (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Generalised oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Early satiety (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypothermia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Irritability (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Localised oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tenderness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 5 | 0 | 2 | 2 | 0 | 7 | 6
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 2 | 6 | 0 | 0 | 2 | 1 | 9 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 0 | 2 | 0 | 0 | 1 | 0 | 5 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 1 | 2 | 0 | 0 | 1 | 0 | 1 | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 4
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cachexia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Iron deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 3 | 3 | 0 | 0 | 3 | 0 | 5 | 3
Headache (Nervous system disorders) | 1 | 0 | 0 | 2 | 0 | 1 | 0 | 2 | 1 | 0 | 0 | 2 | 1 | 2 | 2
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Convulsion (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ataxia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Drug withdrawal headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hemiparesis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperreflexia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Loss of proprioception (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Speech disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vocal cord paralysis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 1 | 2 | 0 | 1 | 1 | 0 | 3 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 3 | 1 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Critical illness myopathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 3 | 0 | 0 | 3 | 0 | 2 | 2
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 0 | 0 | 0 | 1 | 0 | 1
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 4
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Weight increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ammonia increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood potassium decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood pressure increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood urine present (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Carbon dioxide decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Electrocardiogram QRS complex abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haemoglobin (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oxygen saturation decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Platelet count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Protein total decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Waist circumference increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 1 | 0 | 2 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 2 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 3 | 2 | 1
Visual impairment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 3 | 1
Periorbital oedema (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 1 | 0 | 2 | 0
Macular degeneration (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0
Vitreous floaters (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Abnormal sensation in eye (Eye disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ocular icterus (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Uveitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Diplopia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Eye pain (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 1 | 3 | 0 | 0 | 0 | 1 | 3 | 2
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 1
Hordeolum (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Escherichia infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Groin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Herpes virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nail bed infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Peritonitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash pustular (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Syphilis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 2 | 0 | 0 | 0 | 1 | 2 | 1 | 2 | 1 | 0 | 1 | 1 | 0 | 3 | 6
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 0 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Hallucination, visual (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Disorientation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mood swings (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Restlessness (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Procedural site reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Animal bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Incision site pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 2
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 1 | 0
Bloody discharge (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Costovertebral angle tenderness (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nocturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal artery stenosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Scrotal oedema (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Vaginal discharge (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Breast pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Genital rash (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Menstruation irregular (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oedema genital (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vulvovaginal erythema (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Jaundice (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Wisdom teeth removal (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.